CLINICAL TRIAL: NCT03619616
Title: A Phase 1 Randomized,Double-Blind,Parallel-Group, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ZSP1603 in Chinese Healthy Subjects
Brief Title: Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending Dose of ZSP1603 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Zhongsheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XY3-PK-ZSP1603
Record Dates: First submitted 2018-07-23; First posted 2018-08-08 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Idiopathic Pulmonary Fibrosis(IPF); Solid Tumor
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple(Participant, Investigator, Clinical Research Associate)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ZSP1603 (single dose)-7.5 mg (Cohort 1) (Experimental): Subject adminsitered at a dose of ZSP1603 7.5 mg on day 1 under fasted condition.
  Interventions: Drug: ZSP1603 7.5 mg
- ZSP1603 (single dose)-12.5mg (Cohort 2) (Experimental): Subject adminsitered at a dose of ZSP1603 12.5 mg or placebo on day 1 under fasted condition.
  Enrollment into Cohort 2 will begin upon assurance of safety for Cohort 1.
  Interventions: Drug: ZSP1603 12.5 mg; Drug: Placebo 12.5mg
- ZSP1603 (single dose)-25 mg (Cohort 3) (Experimental): Subject adminsitered at a dose of ZSP1603 25 mg or placebo on day 1 under fasted condition.
  Enrollment into Cohort 3 will begin upon assurance of safety for Cohort 2.
  Interventions: Drug: ZSP1603 25 mg; Drug: Placebo 25mg
- ZSP1603 (single dose)-50 mg (Cohort 4) (Experimental): Subject adminsitered at a dose of ZSP1603 50 mg or placebo on day 1 under fasted condition.
  Enrollment into Cohort 4 will begin upon assurance of safety for Cohort 3.
  Interventions: Drug: ZSP1603 50 mg; Drug: Placebo 50mg

INTERVENTIONS:
Drug: ZSP1603 7.5 mg — ZSP1603 capsule administered orally once daily under fasted condition.
  Arms: ZSP1603 (single dose)-7.5 mg (Cohort 1)
Drug: ZSP1603 12.5 mg — ZSP1603 capsule administered orally once daily in the fasting state.
  Arms: ZSP1603 (single dose)-12.5mg (Cohort 2)
Drug: Placebo 12.5mg — Participants will receive placebo matching to ZSP1603 orally once daily under fasted condition.
  Arms: ZSP1603 (single dose)-12.5mg (Cohort 2)
Drug: ZSP1603 25 mg — ZSP1603 capsule administered orally once daily under fasted condition.
  Arms: ZSP1603 (single dose)-25 mg (Cohort 3)
Drug: Placebo 25mg — Participants will receive placebo matching to ZSP1603 orally once daily in the fasting state.
  Arms: ZSP1603 (single dose)-25 mg (Cohort 3)
Drug: ZSP1603 50 mg — ZSP1603 capsule administered orally once daily under fasted state.
  Arms: ZSP1603 (single dose)-50 mg (Cohort 4)
Drug: Placebo 50mg — Participants will receive placebo matching to ZSP1603 orally once daily in the fasting state.
  Arms: ZSP1603 (single dose)-50 mg (Cohort 4)

SUMMARY:
The Primary objectives of this study are to evaluate the safety and tolerability of ZSP1603 and the Secondary objective is to estimate the pharmacokinetic (PK) parameters after orally administered once daily of ZSP1603.

DETAILED DESCRIPTION:
This is a Phase 1, double-blinded, placebo-controlled, single center study aimed at investigating the safety, tolerability and the pharmacokinetics of ZSP1603 on fasted condition.Up to 4 cohorts of 32 eligible participants totally are planned to be enrolled. This is a two-arm clinical trial that ZSP1603 and matching placebo will be orally administered once daily. Two subjects in the first cohort will be assigned in a opened fashion to receive 7.5mg of ZSP1603 while another three cohorts of volunteers will be randomly assigned in a blinded fashion to receive either a single dose of ZSP1603 or matching placebo in an ascending dose fashion. To monitor AEs,record abnormalities (Holter, 12-lead ECG, Vital signs, Physical examination, Clinical Laboratory), and detect the pharmacokinetics of ZSP1603.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are required to meet the following criteria in order to be included in the trial:

  1. Males and female subjects between 18-50 years (Both inclusive).
  2. Body weight is no less than 50 kg in males and no less than 45 kg in females. Body mass index (BMI) 19.0 ≤ BMI ≤ 26.0 kg/m2; BMI is determined by the following equation: BMI = weight/height2 (kg/m2).
  3. Males or females are without gestation plans or infertility, or females who are menopausal, otherwise must use reliable methods of contraception during the study and until 6 months following the last dose of investigational product.
  4. Signature of a dated Informed Consent Form (ICF) indicating that the subject has been informed of all the relevant aspects(including adverse events) of the trial prior to enrollment.
  5. Subjects must be willing and able to adhere to the visit schedule and protocol requirements and be available to complete the study.

Exclusion Criteria:

* Eligible subjects must not meet any of the following exclusion criteria:

  1. History or presence of any clinical severe diseases (such as circulatory system, endocrine , neurologic, gastrointestinal, respiratory system, urogenital system, hematic, immune, psychiatric and metabolic abnormalities), or any other diseases that,in the Investigator's opinion,might interfere with the assessment or follow-up;
  2. Known hypersensitivity and/or allergy to some drugs and food,especially for the composition that is similar to the investigative product;
  3. Subjects who have received a surgery within 4 weeks prior to the test or who plan to perform a surgery during the study;
  4. Use of any drugs or health care products (including herbs) within 14 days prior to screening.
  5. Any drugs with known hepatic enzyme-inducing or inhibiting agents that may change the activity of CYP3A4 within 30 days prior to dosing (such as inducer - Barbituric , Carmazepin , Phenyltoin , Glucocorticoids , and Omeprazole ; Inhibitors - SSRI antidepressants , Cimitedin , Diltiazem , Macrolides , Nitroimidazoles , Sedative hypnotic , Verapamil , Fluoroquinolone , Anti - histamine ).
  6. Participated in another clinical research study and received any other investigational products within 3 months prior to dosing.
  7. Subjects who donated blood or bleeding profusely(≥ 200 mL), received blood transfusion or use of blood products in the 3 months preceding study screening.
  8. Pregnancy or breastfeeding at screening and during the study. All female subjects of childbearing potential and their partners cannot use at least one reliable method of non-drug contraception during the study and until 6 months following the last dose of investigational product.
  9. Subjects who have special dietary habit and inability to consume the food provided in the study;
  10. Subjects who could not tolerate venipuncture;
  11. Dysphagia of capsule;
  12. Frequently drinks tea, coffee and/or caffeinated beverages(more than 8 cups, 1 cup =250 mL) per day ;
  13. Daily consuming more than 5 cigarettes within 3 months prior to screening or cannot stop using any tobacco products during the trial.
  14. Smoke or have grapefruit juice,any food or beverage that contains alcohol or xanthin (including chocolate, tea, coffee, cola, etc.) from 48 hours pre-dose to the last blood collection ;
  15. Known history of alcohol abuse (defined as consumption of more than 14 units of alcohol per week: 1 unit=360 ml of beer,or the equivalent of 45 mL liquor with 40% alcohol content, or 150 ml of wine;)or take any product contains alcohol during the study.
  16. Known history of drug abuse or subjects who have used soft drugs (e.g., marijuana) within 3 months prior to screening, or have taken hard drugs (such as cocaine, phencyclidine, etc.) within one year before screening.
  17. Presence clinically significant abnormalities (based on the judgment of clinical research doctors) of vital signs (systolic pressure <90 mmHg or >140 mmHg; diastolic pressure <60 mmHg or >90 mmHg；HR <50 bpm or>100 bpm) or ECG (QTcB>450ms in males, or QTcB>480ms in females) or physical examination, clinical laboratory tests and imaging examination.
  18. Subjects who may not complete the study for other reasons or should not be included in the study in the opinion of the Investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) following oral doses of ZSP1603 and placebo,separately. | At Day 6 post-dose.
  Number of participants with TEAEs as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
AUClast（AUC0-t）of ZSP1603 | Up to 6 days post-dose
  AUClast is defined as the concentration of drug from time zero to the last quantifiable concentration.
AUC0-24 of ZSP1603 | Up to 6 days post-dose
  AUC0-24 is defined as the concentration of drug from zero(0) hrs to 24h (area under the plasma concentration versus time curve from zero(0) hrs to 24h).
Cmax of ZSP1603 | Up to 6 days post-dose
  Cmax is defined as the maximum observed concentration of drug in plasma.
Tmax of ZSP1603 | Up to 6 days post-dose
  Tmax is defined as the time to maximum concentration.
t1/2 of ZSP1603 | Up to 6 days post-dose
  t1/2 is defined as the time to half of the drug concentration in plasma.
CL/F of ZSP1603 | Up to 6 days post-dose
  CL/F is defined as the ratio of total clearance(CL) to bioavailability(F).
λz of ZSP1603 | Up to 6 days post-dose
  λz is defined as the ratio between the elimination of compound per unit time and the total amount of compound.
VD/F of ZSP1603 | Up to 6 days post-dose
  VD/F is defined as apparent volume of distribution
MRT of ZSP1603 | Up to 6 days post-dose
  MRT is defined as mean residence time

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Yang, MD, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China